CLINICAL TRIAL: NCT02690168
Title: Testing Glial Pathways to HAAF in Human Subjects Using Carbon 13 Magnetic Resonance Spectroscopy
Acronym: GLIMpSE
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, David McDougal, Assistant Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2015-019
Record Dates: First submitted 2016-01-27; First posted 2016-02-24 (Estimated); Results first posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Complications; Hypoglycemia
Keywords: Fasting; Carbon-13 Magnetic Resonance Spectroscopy; Neuroimaging
MeSH Terms: conditions — Diabetes Complications; Hypoglycemia; Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood banking
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Men
  Interventions: Behavioral: Fasting

INTERVENTIONS:
Behavioral: Fasting — 72 hour fasting

SUMMARY:
Hypoglycemia-associated autonomic failure (HAAF), a condition commonly developed in diabetic patients, which causes them to have severely low blood sugar levels. This condition makes clinical management of blood sugar in diabetic patients very challenging. This research seeks to better understand how diabetic patients develop HAAF, and what can be done to prevent it.

DETAILED DESCRIPTION:
Following the detection of severe hypoglycemia by the central nervous system (CNS), a series of physiological countermeasures are triggered which return serum glucose to euglycemic levels. This vital homeostatic response frequently becomes dysfunctional in both type 1 and type 2 diabetics, leaving them particularly vulnerable to life threatening bouts of hypoglycemia. This dysfunction, often termed hypoglycemia-associated autonomic failure (HAAF), is thought to be caused by maladaptive changes in the CNS. Currently, progress towards rectifying this HAAF is severely hindered by a lack of knowledge regarding the exact nature of these maladaptive changes and the antecedent events which cause them. Previous work by the PI, as well as others, has identified altered glial metabolism as a potential biological substrate driving HAAF. The alterations in glial metabolism associated with HAAF are strikingly similar to those induced by prolonged dietary restriction in rodents. This raises the intriguing possibility that HAAF may be driven by glial adaptations, normally induced only by prolonged starvation, which are triggered in diabetic individuals by treatment-induced exposure to severe hypoglycemia. The primary goal of our pilot project is to conduct a prospective observational study in humans to test the hypothesis that prolonged fasting will induce changes in glial metabolism similar to those previously measured in individuals with HAAF. The investigators will accomplish this goal via the following specific aims: Aim 1: Using a prospective observational study design in humans, test whether a 72 hour fast will induce acute alterations in glial metabolism, Aim 2: Determine if changes in plasma glucose and leptin levels following prolonged fasting are correlated with changes in glial adaptation. The investigators will utilize innovative 13C magnetic resonance spectroscopy to measure alterations in glial metabolism and substrate preference following acute dietary restriction in healthy young individuals. By demonstrating that metabolic adaptations of glial cells induced by prolonged fasting are similar to those previously associated with HAAF, the investigators can provide key insights into the precursors that may lead to the development of HAAF in diabetic individuals.

ELIGIBILITY:
Inclusion Criteria:

* Male
* BMI 20.0-24.9 kg/m2
* 18-40 years old
* Willing to reside at Pennington Biomedical for 4 days

Exclusion Criteria:

* Type 1 diabetes mellitus
* Type 2 diabetes mellitus
* Fasting glucose ≥ 110 mg/dL (determined at screening visit)
* Hyperketonuria >15 mg/dL, (determined at screening visit)
* Contraindication to MRI
* History of or current eating disorder
* History of obsessive compulsive disorder
* Current use of any medication (excluding over-the-counter pain medication)
* Contraindication to prolonged fasting
* Consume >10 alcoholic drinks/week

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Men
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David McDougal, PhD, Principal Investigator — Pennington Biomedical Rsrch Ct
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] McDougal DH, Darpolor MM, DuVall MA, Sutton EF, Morrison CD, Gadde KM, Redman LM, Carmichael OT. Glial acetate metabolism is increased following a 72-h fast in metabolically healthy men and correlates with susceptibility to hypoglycemia. Acta Diabetol. 2018 Oct;55(10):1029-1036. doi: 10.1007/s00592-018-1180-5. Epub 2018 Jun 22. PMID 29931424

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fasting
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Men
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kg] | 76.1 (13.7)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23.5 (2.7)
Fasting glucose [Mean (Standard Deviation); unit: mg/dL] | 85.1 (6.9)
% body fat [Mean (Standard Deviation); unit: % body fat] | 17.6 (7.3)
Percent enrichment of bicarbonate [Mean (Standard Deviation); unit: % enrichment] — Population: Collected data from one participant were not considered valid due to an equipment malfunction
  % enrichment
    number analyzed (Participants) | 5
    (all) | 53.5 (8.3)
Cerebral Metabolic Rate of Acetate Ascertained Through Mathematical Modeling of MRS Data [Mean (Standard Deviation); unit: micromol/g/min] — Population: Collected data from one participant were not considered valid due to an equipment malfunction
  micromol/g/min
    number analyzed (Participants) | 5
    (all) | 59 (20.8)
Astroglial tricarboxylic acid cycle rate ascertained through mathematical modeling of MRS data [Mean (Standard Deviation); unit: micromol/g/min] — Population: Collected data from one participant were not considered valid due to an equipment malfunction
  micromol/g/min
    number analyzed (Participants) | 5
    (all) | 0.5 (0.2)
Leptin [Mean (Standard Deviation); unit: ng/mL] — Population: parameter could only be measured in 3 subject due to lack of collected blood volume
  ng/mL
    number analyzed (Participants) | 3
    (all) | 7.2 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Percent Enrichment of Bicarbonate as Measured by Magnetic Resonance Spectroscopy (MRS)
Time Frame: 80 hours
Population: Collected data from one participant were not considered valid due to an equipment malfunction
Measure: Mean (Standard Deviation); unit: % enrichment
Arm/Group | Healthy Men
Number analyzed (Participants) | 5
% enrichment | 61.9 (3.8)
Statistical Analysis 1: Comparison: Healthy Men; Test type: Other; p = 0.0053, t-test, 2 sided

2. Secondary Outcome: Cerebral Metabolic Rate of Acetate Ascertained Through Mathematical Modeling of MRS Data
Time Frame: 80 hours
Population: Collected data from one participant were not considered valid due to an equipment malfunction
Measure: Mean (Standard Deviation); unit: micromol/g/min
Arm/Group | Fasting
Number analyzed (Participants) | 5
micromol/g/min | 71 (15.0)
Statistical Analysis 1: Comparison: Fasting; Test type: Other; p = 0.477, t-test, 2 sided

3. Secondary Outcome: Astroglial TCA Cycle Rate Ascertained Through Mathematical Modeling of MRS Data
Time Frame: 80 hours
Population: Collected data from one participant were not considered valid due to an equipment malfunction
Measure: Mean (Standard Deviation); unit: micromol/g/min
Arm/Group | Fasting
Number analyzed (Participants) | 5
micromol/g/min | 0.4 (0.2)
Statistical Analysis 1: Comparison: Fasting; Test type: Other; p = 0.917, t-test, 2 sided

4. Secondary Outcome: Glucose Level
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Fasting
Number analyzed (Participants) | 6
mg/dL | 71 (4.9)

5. Secondary Outcome: Change in Leptin Levels
Time Frame: 72 hours
Population: Data from 3 participants was not available due to lack of blood volume during collections
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Fasting
Number analyzed (Participants) | 3
ng/mL | 5.2 (1.2)
Statistical Analysis 1: Comparison: Fasting; Test type: Other; p = 0.53, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 4 days
Arm/Group | Fasting
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fasting (N=6)
Achy legs (Musculoskeletal and connective tissue disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
insomnia (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-22): https://cdn.clinicaltrials.gov/large-docs/68/NCT02690168/Prot_SAP_000.pdf